CLINICAL TRIAL: NCT00583440
Title: 12-step Facilitation for the Dually Diagnosed
Acronym: TSFDD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael Bogenschutz, Professor of Psychiatry, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA-Bogenschutz-AA015419; R01AA015419 (NIH); NIH Grant 1R01 AA015419
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Alcoholism; Diagnosis, Dual (Psychiatry)
Keywords: 12-step; mutual help; dual diagnosis; serious mental illness
MeSH Terms: conditions — Alcoholism; Disease | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: 12-step facilitation
- 2 (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: 12-step facilitation — 12 weekly individual 12-step facilitation sessions
  Arms: 1
Behavioral: Treatment as usual — Usual clinical treatment in a dual diagnosis treatment program
  Arms: 2

SUMMARY:
This is a randomized trial testing the efficacy of a modified 12-step facilitation therapy for individuals with serious mental illness and alcohol use disorders, compared to usual treatment. 135 participants are randomized in 2:1 ratio to the modified 12-step facilitation (12 sessions of individual counseling) vs. treatment as usual. The primary hypothesis is that those receiving 12-step facilitation will have better drinking outcomes (percent days abstinence and drinks per drinking day)at end of treatment.

DETAILED DESCRIPTION:
Although there has been relatively little work on 12-step treatment for seriously mentally ill patients, extant literature indicates that dually diagnosed individuals attend traditional 12-step programs such as AA, NA, and CA at rates comparable to singly diagnosed substance abusers, and that participation is associated with decreases in substance use. Specialized 12-step programs for the dually diagnosed, developed over the past 10 years, may offer additional benefits. In order to maximize the effectiveness of specialized and traditional 12-step programs for dually diagnosed individuals, specially adapted 12-step facilitation (TSF) treatment for the dually diagnosed should be developed and tested. Standard TSF should be modified to address the special needs of dually diagnosed individuals, mesh with specialized 12-step programs available in the area, and address barriers to attendance, participation, and engagement experienced by the dually diagnosed. We have developed a modified TSF based on the Project MATCH TSF manual. Modifications to this 12 week individual therapy include: emphasis on specialized 12-step program attendance; readings primarily from specialized 12-step program literature; participation in the second session by a community specialized 12-step program member; case management to assist participants in finding and attending meetings; omission of work on the fourth step; and the addition of topics covering medication compliance and specific social skills needed to negotiate 12-step meetings. In a pilot study with 10 dually diagnosed individuals, participants showed significant decreases in substance use and significant increases in 12-step attendance after receiving the specialized TSF. Building on this pilot study, the proposed study is a larger Stage 1b study of the modified TSF for seriously mentally ill patients engaged in dual diagnosis treatment. Participants with a psychotic or major affective disorder will be randomized to modified TSF (n=90) vs. treatment as usual (n=45). Participants will be followed for a total of 48 weeks. Assessments will include rigorous diagnosis and measures of alcohol and other drug use, consequences, psychiatric symptoms, 12-step behaviors, 12-step specific and non-specific change mechanisms, and social support. Specific Aims of the study include assessment of the integrity of the planned intervention and assessment battery; tests of the effectiveness of the adapted TSF relative to treatment as usual; determination of whether psychiatric diagnosis moderates treatment response; and investigation of causal mechanisms of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. SCID Diagnosis of a psychotic disorder (schizophrenia, schizoaffective disorder, or psychosis not otherwise specified) or a major affective disorder (major depression, bipolar disorder, or depressive disorder not otherwise specified, provided in the latter case that criteria have been met for a major depressive episode).
2. SCID diagnosis of alcohol abuse or dependence which is active within the past 1 month (i.e., not in early or sustained full remission).
3. Two or more days of heavy drinking (5 or more drinks for per occasion for a man, 4 or more drinks per occasion for a woman) in the 30 days prior to screening.
4. Willingness to participate in specialized 12-step programs.
5. Ability to provide informed consent.
6. Ability to read, speak, and understand English at least the 5th grade level.
7. Ability to provide at least one contact person to assist in tracking for follow-up assessment.

Exclusion Criteria:

1. Current attendance of any 12-step program (two or more 12-step meetings in the past month).
2. Unstable psychiatric illness, defined by psychiatric hospitalization in the past 1 month; more than 3 hospitalizations in the past year; or psychosis or mania which would render the individual incapable of informed consent.
3. Active suicidality (any clinically significant suicide attempts in the past 3 months or any current suicidal intent or definite plan).
4. Current homicidal ideation aimed at a specific person or persons.
5. Medical illness which is severe enough to compromise participation in the study.
6. Mental retardation, dementia, or other cognitive impairment of sufficient severely to render the individual incapable of informed consent or incapable of comprehending and participating in the TSF therapy or 12-step meetings.
7. Expectation of being out of town or in jail for more than 21 days during the treatment period.
8. Expectation of participation in any other formal addiction treatment during the study period (not including TAU, 12-step or other mutual support groups).
9. Current engagement in behavioral health treatment (including case management) at another facility.
10. Current engagement in non-TAU treatment at UNMPC, such as psychotherapy, intensive outpatient treatment, or MET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2005-09; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent from alcohol | 12, 24, 36, and 48 weeks

SECONDARY OUTCOMES:
Drinks per drinking day | 12, 24, 36, and 48 weeks
12-step participation | 12, 24, 36, and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Bogenschutz, MD, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- UNM HSC Department of Psychiatry Clinical Trials, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Houck JM, Forcehimes AA, Gutierrez ET, Bogenschutz MP. Test-retest reliability of self-report measures in a dually diagnosed sample. Subst Use Misuse. 2013 Jan;48(1-2):99-105. doi: 10.3109/10826084.2012.731674. Epub 2012 Oct 25. PMID 23098171